CLINICAL TRIAL: NCT06128941
Title: Influence of Physical Training Protocols in Hypoxic, Normobaric and Hypobaric Environments, on the Immune, Metabolic Response and Cardiopulmonary Behavior in Athletes Convalescent From Covid-19
Brief Title: Influence of Hypoxic, Normobaric and Hypobaric Training on the Immunometabolism of Post-covid-19 Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Collaborators: University of Sao Paulo (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Cristina Monteiro, Assistant professor, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SprintRepHipoxya
Record Dates: First submitted 2023-11-09; First posted 2023-11-13 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Normobaric Hypoxia; Hypoventilation; Normoxia
Keywords: HIF1a; HLA-G; Repeated sprint; Inflammation; covid-19; immune system; athletes
MeSH Terms: conditions — Hypoventilation; Inflammation; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normobaric hypoxia (SRH) (Experimental): Participants will carry out training sessions in a normobaric hypoxia chamber at a simulated altitude of 3000 meters (FiO2 14.5%)
  Interventions: Other: Repeated sprint
- Hypoventilation (SRH-VLH) (Experimental): Participants will be asked to exhale to residual functional capacity, immediately before starting each sprint, and to hold their breath until the end of the sprint
  Interventions: Other: Repeated sprint
- Normoxia (SRN) (Active Comparator): Participants will carry out training sessions in normoxia (FiO2 20.9%)
  Interventions: Other: Repeated sprint

INTERVENTIONS:
Other: Repeated sprint — * Duration of the study: 8 weeks of participation.
  * Each repeated sprint training protocol: 2 training sessions per week for 4 weeks.
  * Collection sessions: 3 collection sessions will be carried out: before the start of the training protocol - T0; at the end of the protocol, in week 4 - T1; and late, 4 weeks after the end of the protocol, in week 8 - T2.
  * Training sessions: will be carried out on an ergometer and will consist of 3 sets of 5 sprints of 10s all-out with 20s of rest between sprints, and 5 minutes of rest between sets.

SUMMARY:
COVID-19 has significantly impacted sports globally, with event postponements, training disruptions, and wide-ranging concerns. SARS-CoV-2 infection can result in hyperinflammation and cardiopulmonary changes, with hypoxia as an aggravating sign. Hypoxia triggers complex immunometabolic mechanisms, including activation of HIF-1α and induction of HLA-G expression. Hypoxia training protocols benefit aerobic capacity and sports performance, with potential immunological impact. Studying immunometabolic markers in this context can improve athletic preparation and athletes' general health.

DETAILED DESCRIPTION:
Covid-19, caused by SARS-CoV-2, can progress to pulmonary hyperinflammation and cardiopulmonary changes, with hypoxia being one of the main signs of worsening. In hypoxia, there is activation of HIF-1 that induces the expression of HLA-G, an immuno-tolerogenic molecule that inhibits the hyperinflammatory response. Hypoxia training protocols can promote cardiopulmonary benefits and increase the expression of anti-inflammatory cytokines, HIF-1 and HLA-G. Immunometabolic markers have the potential to be used in the prevention, diagnosis, and treatment of diseases with inflammatory mechanisms. The objective of this study is to evaluate the influence of physical training protocols in hypoxic, normobaric, and hypobaric environments, on the immune, and metabolic response and cardiopulmonary behavior in athletes post covid-19, to identify potential biomarkers and better clarify the impact of exercise on immunometabolism post-covid-19. The study will consist of a randomized and controlled intervention, with training using different normobaric hypoxic methods; and an observational study at natural altitude (hypobaric hypoxia). In the normobaric hypoxia trial, participants will be divided into a control group that will carry out a training plan of repeated sprints in normoxia; and two other groups that will perform the same training sessions in normobaric hypoxia and with low lung volume voluntary hypoventilation. In the observational study with hypobaric hypoxia, high-performance resistance athletes will be recruited, who will comply with the training plan proposed by the team's coach at altitude. Cardiorespiratory, immunometabolic, neuromuscular, and autonomic fatigue, hematological indicators, plasma levels of lipid mediators, sHLA-G and cytokines, and the expression of HIF-1α in leukocyte cells will be evaluated. The analysis of the effect of the training methods will be carried out by ANOVA for repeated measures (parametric or non-parametric), or means comparison tests for paired samples (t or Wilcoxon) after evaluating the assumptions and the identification of associations between variables will be carried out by Binomial Logistic Regression Analysis.

ELIGIBILITY:
Inclusion Criteria:

* more than 5 years of training experience in an resistance modality;
* participates in national or international championships regularly;
* athletes convalescing from covid-19, at least 30 days after diagnosis and/or hospital discharge;
* manifested mild to severe symptoms;
* vaccinated or not against SARS-CoV-2;
* antigen self-test for SARS-CoV-2 negative.

Exclusion Criteria:

* athletes who have had an acclimatization experience or exposure to altitude lasting more than 10 days in the last 6 months;
* contain signs or symptoms of acute covid-19;
* present a positive SARS-CoV-2 antigen self-test;
* pregnant or postpartum women;
* use anti-inflammatory or immunosuppressive medications.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Hypoxia Inducible Factor 1 alpha (HIF-1a) | Before, just after and 4 weeks after the training program
  Flow cytometry for PBMCs
Human Leukocyte Antigen-G (HLA-G) | Before, just after and 4 weeks after the training program
  ELISA
Cytokines (TNF-α, IL-1β, IL-6, IL-10, IL-8 and IFN-γ) | Before, just after and 4 weeks after the training program
  ELISA
Plasma levels of eicosanoids, endocannabinoids, steroid hormones, sphingolipids, ceramides and other glycerophospholipids | Before, just after and 4 weeks after the training program
  Mass Spectrometry (LC-MS/MS)
Hematological indicators (hematocrit, hemoglobin and cell count) | Before, just after and 4 weeks after the training program
  Blood count
Ventilatory thresholds and maximum oxygen consumption | Before, just after and 4 weeks after the training program
  mL/kg·min
Blood lactate concentrations | Before, just after and 4 weeks after the training program
  mmol.L-1
Muscle oximetry | Before, just after and 4 weeks after the training program
  Near-infrared spectroscopy (NIRS)
Peak force | Before, just after and 4 weeks after the training program
  Isometric mid thigh pull

SECONDARY OUTCOMES:
Heart rate | Throughout the training program, 4 weeks
  maximum values during the training sessions (bpm)
Arterial oxygen saturation | Throughout the training program, 4 weeks
  oxymetry (%)
Subjective perception of effort | Throughout the training program, 4 weeks
  Adapted Borg scale
Blood pressure, heart rate and temperature | Before, just after and 4 weeks after the training program
  Values at rest mmHg, bpm and ºC
Anthropometric assessments and body composition | Before, just after and 4 weeks after the training program
  height (m), body mass (kg), fat free mass (kg), fat mass (kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Human Kinetics, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No